CLINICAL TRIAL: NCT00859729
Title: DNA Vaccine Coding for the Rhesus Prostate Specific Antigen (rhPSA) and Electroporation in Patients With Relapsed Prostate Cancer. A Phase I/II Study
Brief Title: Dose Finding Study of a DNA Vaccine Delivered With Intradermal Electroporation in Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Karolinska Institutet (Other); Cyto Pulse Sciences, Inc. (Industry)
Responsible Party: Principal Investigator, Jeffrey Yachnin, Prinicple Investigator, Uppsala University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pVAX/rhPSA -EP 2006; EudraCT # 2006-001128-38
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Prostate Cancer
Keywords: DNA; Vaccine; Electroporation; xenogenic; PSA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort I (Experimental): 50 µg DNA/dose, 3 patients
  Interventions: Biological: pVAXrcPSAv53l (DNA encoding rhesus PSA); Device: DERMA VAX™ intradermal DNA delivery system
- Cohort II (Experimental): 150 µg DNA/dose, 3 patients
  Interventions: Biological: pVAXrcPSAv53l (DNA encoding rhesus PSA); Device: DERMA VAX™ intradermal DNA delivery system
- Cohort III (Experimental): 400 µg DNA/dose, 3 patients
  Interventions: Biological: pVAXrcPSAv53l (DNA encoding rhesus PSA); Device: DERMA VAX™ intradermal DNA delivery system
- Cohort IV (Experimental): 1000 µg DNA/dose, 3 patients
  Interventions: Biological: pVAXrcPSAv53l (DNA encoding rhesus PSA); Device: DERMA VAX™ intradermal DNA delivery system
- Cohort V (Experimental): Optimal dose to be determined, 6 patients
  Interventions: Biological: pVAXrcPSAv53l (DNA encoding rhesus PSA); Device: DERMA VAX™ intradermal DNA delivery system

INTERVENTIONS:
Biological: pVAXrcPSAv53l (DNA encoding rhesus PSA) — 5 doses, 4 weeks apart
  Other Names: rhPSA
Device: DERMA VAX™ intradermal DNA delivery system — in vivo electroporation is applied after each DNA injection
  Other Names: Derma Vax

SUMMARY:
This study will assess the feasibility and safety of vaccination with increasing doses of xenogenic DNA administered intradermally in combination with electroporation in patients with relapse of prostate cancer. The DNA encodes prostate specific antigen (PSA) from Rhesus Macaque (Macaca mulatta), a protein that is 89% homologous to human PSA. The study will also assess the safety and functionality of the DERMA VAX™ (Cyto Pulse Sciences) DNA vaccine delivery system.

ELIGIBILITY:
Inclusion Criteria:

* Male patients. Age >18 years.
* HLA-A*0201 positive.
* Histologically confirmed prostate cancer.
* Minimum two (2) and maximum four (4) years after treatment with curative or salvage radiotherapy.
* Serum testosterone within normal range.
* Increasing PSA from a previous reference value on two (2) consecutive occasions at least one month apart and with a minimum of 2 ng/mL above nadir.
* PSA doubling time is one (1) year or less.
* No evidence of metastatic prostate cancer.
* Karnofsky performance status ≥ 80.
* Adequate organ function:

  * AST and ALT ≤ 2.0 x upper limit of normal (ULN); total serum bilirubin ≤ 1.5 x ULN
  * Calcium ≤ 2.6 mmol/L, serum creatinine ≤ 1.5 x ULN
  * Hb ≥ 100 g/L; absolute leukocyte count ≥ 3.0 x 109 /L; platelets ≥100 x 109 /L
* Life expectancy ≥ 12 months.
* Swedish or English speaking subjects only.
* Written informed consent (subjects must be capable of providing their own informed consent).

Exclusion Criteria:

* Previous ablation of testis.
* Radiologic evidence of metastatic disease.
* Prior chemotherapy or investigational therapy/agents within 4 weeks.
* Active bacterial, viral or fungal infection.
* Carrier of HIV, HBV, or HCV.
* Immunosuppressed (post splenectomy, post stem cell transplantation) or on immunosuppressive therapy other than inhaled or replacement corticosteroids.
* Any other major illness or peripheral blood vein status that, in the investigator's judgement, will substantially increase the risk associated with sampling or participation in this study.
* Subjects with cardiac demand pacemakers.
* Any reason why, in the opinion of the investigator, the patient should not participate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Assess the feasibility and safety of escalating doses of pVAXrcPSAv53l DNA vaccine, administered intradermally in combination with electroporation in patients with relapse of prostate cancer. | From start of treatment to 30 days (safety) or up to 12 months (immunological & clinical) post last vaccination

SECONDARY OUTCOMES:
Assess the safety and functionality of the DERMA VAX™ in vivo electroporation DNA vaccine delivery system. | From start of treatment to 30 days (safety) or up to 12 months (immunological & clinical) post last vaccination
Evaluate the PSA-specific immune response induced by the vaccine. | From start of treatment to 30 days (safety) or up to 12 months (immunological & clinical) post last vaccination
Identify an anti-tumor effect of the vaccine. | From start of treatment to 30 days (safety) or up to 12 months (immunological & clinical) post last vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Yachnin, MD, PhD, Principal Investigator — Department of Oncology, University Hospital Uppsala
Locations (1):
- Department of Oncology, University Hospital Uppsala, Uppsala, Sweden